CLINICAL TRIAL: NCT04680468
Title: Phase 2 Study of Belantamab Mafodotin as Pre- and Post-autologous Stem Cell Transplant Consolidation and Maintenance for Multiple Myeloma
Brief Title: Study of Belantamab Mafodotin as Pre- and Post-autologous Stem Cell Transplant and Maintenance for Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 37420; IRB#844252 (Other: University of Pennsylvania)
Record Dates: First submitted 2020-12-02; First posted 2020-12-23 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Belantamab mafodotin (Experimental): Patients receive Belantamab mafodotin 2.5 mg/kg by intravenous infusion on day -42 relative to autologous stem cell infusion (day 0), on day +60, and every 90 days thereafter, for up to 2 years following ASCT.
  Interventions: Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Belantamab mafodotin — 2.5 mg/kg IV
  Other Names: GSK2857916

SUMMARY:
This is a single-institution, single-arm, phase 2 study in which belantamab mafodotin (GSK2857916), an antibody-drug conjugate targeting B-cell maturation antigen (BCMA), will be administered to patients with multiple myeloma prior to and following high-dose melphalan and autologous stem cell transplantation (ASCT), in conjunction with standard lenalidomide maintenance. We hypothesize that administration of belantamab mafodotin as part of autologous stem cell transplant consolidation and maintenance will be safe, well tolerated, and efficacious in comparison to historical data.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand the study procedures and have signed written, informed consent.
2. Must be 18 years of age or older at enrollment.
3. Must have started therapy for active multiple myeloma within 12 months of enrollment.
4. Must have an ECOG performance status of 0-2.
5. Have received no more than 2 prior lines of induction therapy (induction regimen not specified by protocol), with no prior progressive disease by International Myeloma Working Group (IMWG) criteria.
6. Must be in at least a partial response (PR) but not in a complete response (CR) or better after at least 4 cycles of induction therapy, per IMWG consensus criteria.
7. Eligible by institutional criteria to receive melphalan at a dose of 200 mg/m2.
8. Eligible to receive lenalidomide maintenance therapy post-ASCT.
9. Adequate bone marrow and organ function at enrollment.
10. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

    1. Is not a woman of childbearing potential (WOCBP), OR
    2. Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency, during the intervention period and for at least 4 months after the last dose of belantamab mafodotin and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period.
11. Male participants are eligible to participate if they agree to the following during belantamab mafodotin treatment and for 6 months after the last dose of belantamab mafodotin to allow for clearance of any altered sperm:

    1. Refrain from donating sperm PLUS either:
    2. Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent, OR Must agree to use contraception/barrier as detailed in the protocol.
12. All prior treatment-related toxicities must be grade 1 or less at the time of enrollment except for alopecia.

Exclusion Criteria:

1. Must not have used an investigational drug or approved systemic anti-myeloma therapy (including systemic steroids) within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug.
2. Must not have received treatment with a monoclonal antibody within 28 days of receiving the first dose of study drug
3. Must not be simultaneously enrolled in any interventional clinical trial
4. Must not have amyloidosis or POEMS syndrome.
5. Must not be pregnant or lactating.
6. Must not have current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, severe hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria.
7. Must not have any evidence of active mucosal or internal bleeding
8. History of an active renal condition (infection, requirement for dialysis or any other condition that could affect subject's safety). Subjects with isolated proteinuria resulting from MM are eligible, provided they fulfill other criteria.
9. Participant must not have evidence of cardiovascular risk, as defined in the protocol.
10. Must not have any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormalities) that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
11. Must not have invasive malignancies other than disease under study, unless the second malignancy has been definitively treated or has been medically stable for at least 2 years and, in the opinion of the principal investigator, will not affect the evaluation of the effects of clinical trial treatment.
12. Must not have an active infection requiring antibiotic treatment.
13. Any major surgery within the last 4 weeks prior to enrollment.
14. Must not have current corneal epithelial disease except mild changes in corneal epithelium
15. Must not have known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment
16. Must not have evidence for active hepatitis B infection (i.e. positive hepatitis B surface antigen or nucleic acid-based testing) at screening or within 3 months prior to first dose of belantamab mafodotin.
17. Must not have positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment.
18. Must not have evidence of active HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2026-07-11 (Estimated); Study Completion 2026-07-11 (Estimated)

PRIMARY OUTCOMES:
MRD (minimal residual disease) negativity rate | 12 months post-ASCT
  Percentage of participants who have achieved minimal residual disease (MRD) negativity by next-generation sequencing (NGS) at 12 months post-autologous stem cell transplant (ASCT)

SECONDARY OUTCOMES:
Frequency of treatment-related adverse events | through study completion, approximately 3 years
  Percentage of participants who develop adverse and serious adverse events, including ocular adverse events.
Dose reductions | through study completion, approximately 3 years
  The percentage of participants who require reduction of the dose of belantamab mafodotin will be assessed
Dose delays | through study completion, approximately 3 years
  The percentage of participants who require a delay in dosing of belantamab mafodotin will be assessed
MRD Negativity Rate | at 3 and 24 months post-ASCT
  Percentage of participants who have achieved minimal residual disease (MRD) negativity by next-generation sequencing (NGS) at 3 and 24 months post-autologous stem cell transplant (ASCT)
Overall response rate | through study completion, approximately 3 years
  Percentage of participants who achieve partial response (PR) or better, as assessed by International Myeloma Working Group (IMWG) criteria.
Very good partial response (VGPR) or better rate | through study completion, approximately 3 years
  Percentage of participants who achieve VGPR or better, as assessed by IMWG criteria.
Complete response (CR) or better rate | through study completion, approximately 3 years
  Percentage of participants who achieve CR or stringent CR, as assessed by IMWG criteria.
Progression-free survival | through study completion, approximately 3 years
  Time from enrollment until progression of disease by IMWG criteria, or death, whichever occurs first
Overall survival | through study completion, approximately 3 years
  Time from enrollment until death from any cause
Stem cell yield | Following stem cell mobilization, about 6 weeks after enrollment
  The number of days required to collect sufficient autologous peripheral blood stem cells to proceed to ASCT will be assessed
Stem cell collection days | Following stem cell mobilization, about 6 weeks after enrollment
  : The number of days required to collect sufficient autologous peripheral blood stem cells to proceed to ASCT will be assessed
Hematopoietic reconstitution post-ASCT | up to 30 days post-ASCT
  The number of days until neutrophil and platelet recovery post-ASCT (defined as absolute neutrophil count >1000 cells/mcl and platelet count >50000 cells/mcl, respectively) will be assessed
Change from Baseline in Health-related quality of life (HRQoL) as assessed by Functional Assessment of Cancer Therapy - Multiple Myeloma (FACT-MM) questionnaire | baseline through study completion, approximately 3 years.
  The FACT-MM questionnaire is a 41 item questionnaire measuring physical, social/family, emotional, and functional well-being, as well as additional concerns

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cohen, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No